CLINICAL TRIAL: NCT05038267
Title: Femoral Venous Pulsatility and Right Heart Dysfunction in Heart Surgery: An Observational Study
Acronym: FemousTechno6
Status: Completed | Type: Observational
Sponsor: Montreal Heart Institute (Other)
Collaborators: Olivier Lachance, MD (Unknown); Melissa Parent, MD (Unknown); Patrick Tawil, MD (Unknown); Etienne Couture, MD PhD (Unknown); William Beaubien Souligny, MD PhD (Unknown); Yoan Lamarche, MD PhD (Unknown); Alexander Calderone (Unknown); Stephanie Jarry, MSc (Unknown); Ali Hammoud, RN (Unknown); Pierre Robillard, MD (Unknown); Olivier Royer, MD (Unknown); Elena Saade, MD (Unknown)
Responsible Party: Principal Investigator, Andre Denault, MD, PhD, FRCPC, ABIM-CCM, Montreal Heart Institute
Other Study IDs: ICM # 2021-2963
Record Dates: First submitted 2021-08-28; First posted 2021-09-09 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Heart; Dysfunction Postoperative, Cardiac Surgery; Right Heart Failure; Right Ventricular Dysfunction
Keywords: Pulsatile Femoral Vein Doppler Flow
MeSH Terms: conditions — Heart Failure; Ventricular Dysfunction, Right

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Femous patients: Adults undergoing general anesthesia for an elective cardiac surgery requiring cardiopulmonary bypass

SUMMARY:
Right heart failure during cardiac surgery is associated with increased perioperative morbidity and mortality. In this context, it is imperative to develop simple diagnostic tools to detect right heart failure. The purpose of this observational study is to determine if ultrasound Doppler of the femoral vein can detect and predict right ventricular failure after cardiac surgeries requiring cardiopulmonary bypass. It is expected that an elevated pulsatility of the femoral vein before the induction of general anesthesia is associated with perioperative right heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Adults (at least 18 years old)
* Able to consent
* Undergoing elective cardiac surgery at the Montreal Heart Institute
* Surgery requiring cardiopulmonary bypass
* Peri-operative trans-oesophageal echography planned

Exclusion Criteria:

* Critical preoperative state, defined as vasopressor requirement, mechanical support including intra-aortic balloon, mechanical ventilation or cardiac arrest necessitating resuscitation
* Know condition that could interfere with femoral venous assessment or interpretation (such as femoral vein thrombosis, femoral instrumentation, ECMO, etc.)
* Planned cardiac transplantation, implantation of a ventricular assist device or surgery for a congenital condition
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults undergoing elective cardiac surgery at the Montreal Heart Institute which requires cardiopulmonary bypass and perioperative trans oesophageal echography
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2021-08-30 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Determine the prevalence of an elevated pulsatility of the femoral vein on Doppler ultrasound before the induction of general anesthesia | Before induction of anesthesia to day 1 postoperatively at the intensive care unit
  An elevated pulsatility on Doppler ultrasound is defined as a biphasic signal of the femoral vein with a retrograde velocity > 10 cm/s on a long axis view at an angle correction < 60 degrees. If there's signs of cardiac modulation on the Doppler ultrasound, pulsatility index will be measured in long and short axis as followed : (maximal velocity - minimal velocity)/maximal velocity.

SECONDARY OUTCOMES:
Determine the association between an elevated femoral vein pulsatility and diastolic or systolic right ventricular failure, before and after cardiac surgery and at the intensive care unit | Before induction of anesthesia to day 1 postoperatively at the intensive care unit
Determine the association between an elevated femoral vein pulsatility and the intracardiac pressures of the right heart cavities and the pulmonary artery | Before induction of anesthesia to day 1 postoperatively at the intensive care unit
Determine the association between the prevalence of an elevated femoral vein pulsatility and the portal vein pulsatility | Before induction of anesthesia to day 1 postoperatively at the intensive care unit
Determine the impact of positive-pressure ventilation on the femoral vein pulsatility | After induction of anesthesia and before cardiopulmonary bypass.
Determine the association between a preoperative elevated femoral vein pulsatility and postoperative complications. | Immediate postoperative to Day 1 postoperatively at the intensive care unit
  Postoperative complications will be defined as prolonged mechanical ventilation, inotropes or vasopressors dependencies, surgical second-look, acute kidney injury, mortality, hemorrhage, surgical sites infections, delirium and strokes
Compare right and left femoral vein Doppler's ultrasound | Before induction of anesthesia to day 1 postoperatively at the intensive care unit
Determine the most valid measure between long and short axis ultrasound of the femoral vein, and their respective sensibility and specificity to predict complications | Before induction of anesthesia to day 1 postoperatively at the intensive care unit
Determine the sensibility and specificity of the values obtained by the femoral vein Doppler ultrasound to predict postoperative complications | Before induction of anesthesia to day 1 postoperatively at the intensive care unit
Determine if the diameter of the femoral vein as a useful predictor of right heart failure or of post-operative complications | Before induction of anesthesia to day 1 postoperatively at the intensive care unit
Determine the association between an elevated femoral vein pulsatility and postoperative delirium (as evaluated by the Intensive Care Delirium Screening Checklist) | Before induction of anesthesia to day 1 postoperatively at the intensive care unit

CONTACTS AND LOCATIONS:
Locations (1):
- Montreal Heart Institute, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hammoud A, Mailhot T, Parent M, Huard K, Lachance O, Tawil P, Calderone A, Levesque S, Jarry S, Beaubien-Souligny W, Couture EJ, Denault AY. Femoral Vein Pulsatility and Neurocognitive Disorder in Cardiac Surgery. CJC Open. 2024 Nov 8;7(2):187-192. doi: 10.1016/j.cjco.2024.11.002. eCollection 2025 Feb. PMID 40060204
- [Derived] Huard K, Lachance O, Parent M, Tawil P, Saade E, Hammoud A, Couture EJ, Lamarche Y, Jarry S, Calderone A, Robillard P, Levesque S, Beaubien-Souligny W, Denault AY. Prevalence of abnormal common femoral vein pulsatility on Doppler ultrasound in patients undergoing cardiac surgery and its association with adverse events: a prospective cohort study. Can J Anaesth. 2025 Apr;72(4):615-626. doi: 10.1007/s12630-025-02911-9. Epub 2025 Mar 3. PMID 40032766
- [Derived] Couture EJ, Gronlykke L, Denault AY. New developments in the understanding of right ventricular function in acute care. Curr Opin Crit Care. 2022 Jun 1;28(3):331-339. doi: 10.1097/MCC.0000000000000946. PMID 35653255